CLINICAL TRIAL: NCT06118801
Title: The Effect of Probiotics Added to the Mother's Diet on the Occurrence of Necrotizing Enterocolitis and Sepsis and Other Parameters in Preterm Babies
Brief Title: The Effect of Probiotics Added to the Mother's Diet on Preterm Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harran University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Filiz Solmaz, lecturer, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HarrranU-FSolmaz-001
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Preterm; Necrotizing Enterocolitis; Late-Onset Neonatal Sepsis; Breast Milk Expression
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing; Neonatal Sepsis; Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Mothers of premature babies in this group will be given breast milk and breastfeeding training immediately after birth in order to ensure that they can give only breast milk to their babies, and at the same time, 80 ml of probiotic supplements will be given once a day for 20 days.
  Interventions: Dietary Supplement: Probiotic Product Supplement
- control group (No Intervention): There will be no intervention for mothers of preterm babies in this group, and they will be trained on breast milk and breastfeeding so that they can give only breast milk to the baby.

INTERVENTIONS:
Dietary Supplement: Probiotic Product Supplement — Mothers of preterm babies who feed their babies only with breast milk will be given a probiotic product supplement once a day (80 ml probiotic product support containing the Actregularis (5×106 CFU\mL) (lactobacillus bulgaricus, streptococcus thermophilus, lactococcus lactis and bifidobacterium lactis) strain)
  Arms: Probiotic group

SUMMARY:
Abstract According to the definition by World Health Organization; births before the completion of the 37th gestational week are called, preterm birth. Preterm birth is among the most important causes of mortality and morbidity during infancy. Necrotizing enterocolitis (NEC) is the most common gastrointestinal emergency encountered in the Neonatal Intensive Care Unit. The most common risk factors are, preterm birth, enteral feeding and bacterial colonization.

Late Onset Sepsis (LOS) is one of the most common causes of morbidity and mortality in the preterm infants. A healthy gut microbiota has a key role in developing and maintaining a balanced immune response and establishing the intestinal barrier in the immediate postnatal period. Probiotics come to the fore as means that may be effective in preventing NEC and LOS.

Although it is widely accepted that, breast milk has its own microbiota, the origin of these bacterial populations in the milk, has not been fully understood. The new information regarding especially the anaerobic species associated with the intestinal environments that cannot be found in the aerobic environments, suggests an endogenous route to the mammary gland through the presence of the entero-mammary pathway.

The aim of this project is to determine the effect of the probiotics added to the maternal diet on the incidence of encountering NEC and LOS in the preterm infants. The unique value of this project is that, 80 ml of probiotic yogurt will be given to mothers of the preterm infants, who still breastfeed their babies, for 20 days and the effects on the baby will be examined in the scope of the study.

The study has been planned to be conducted as a randomized controlled study in the Neonatal Intensive Care Unit of Şanlıurfa Training and Research Hospital. The power analysis was performed with G*Power for the sample size of the study, which has an experimental/control design structure. The sample size was determined as 50 in total. Data collection tools were organized as Mother and Infant Introductory Information Form (23 questions), Mother and Infant Follow-up Form during Probiotic Implementation (7 questions). At the beginning of the study, all mothers will fill out the mother and baby introductory information form, and the mothers in the experimental group will be given 80 ml probiotic yogurt support once a day for 20 days. In addition to that, all the babies will be monitored for growth once a week, throughout the process. Their status of regular breastfeeding, whether they are diagnosed with NEC and LOS, the time of transition to oral feeding, their bilirubin levels, their status of receiving phototherapy and their discharge durations will be evaluated, and a questionnaire that consists of scale questions will be applied after the discharge.

As a result of this project, it is aimed with the probiotic that will be added to maternal nutrition to reduce the encounter of NEC and LOS in preterm infants, to positively affect the intestinal microbiota by preventing dysbiosis in these infants, to protect them from very important problems such as NEC and LOS as well as accelerating the transition to oral feeding, to help them gain weight, to shorten the duration of receiving phototherapy and hospitalization by reducing the bilirubin levels.

DETAILED DESCRIPTION:
Preterm birth is birth that occurs before the completion of the 37th week of pregnancy. It affects approximately 10% of pregnancies and is a leading cause of perinatal morbidity and mortality. Preterm infants are at high risk for necrotizing enterocolitis (NEC), sepsis, death, and lifelong neurodevelopmental and cognitive impairment.

The most important acquired disease of the gastrointestinal tract in preterm infants is NEC, which is characterized by intestinal necrosis of varying depths and locations and most commonly affects the terminal ileum and proximal colon. NEC is a devastating disease with multifactorial etiology that carries a great burden in terms of mortality, morbidity, and cost to society. It is seen with a frequency of 3-15% in neonatal intensive care units, and >90% of affected babies are preterm babies under 32 weeks of gestation . According to the data of the Turkish Neonatology Association, the incidence in very low birth weight (VLBW) babies is 9.1% . Although its etiology and pathogenesis are not fully understood, it is a condition characterized by inflammation-related ischemic necrosis of the intestinal mucosa. Despite early diagnosis and aggressive treatment, it causes 15-30% mortality and is an important cause of long-term morbidity, especially in VLBW babies. The inflammatory process initiated in the highly immunoreactive gut in NEC prolongs the effects of the disease systemically, affecting distant organs such as the brain and placing affected infants at significantly increased risk for neurodevelopmental delays . One hypothesis suggests that the main etiological factor for NEC is colonization of the neonatal intestine with an abnormal microbiota, specifically that NEC typically occurs 8-10 days after birth when anaerobic bacteria begin to colonize the intestine. In studies examining the effectiveness of probiotic supplementation in preventing NEC (Evidence Level 1+, Recommendation Level B/C), there was a significant reduction in overall mortality. concluded Neonatal sepsis is a clinical syndrome in which there are systemic signs and symptoms of infection in the first month of life and a specific agent is produced in blood culture. Despite the developments in the field of neonatology, it is still an important cause of morbidity and mortality. The incidence of neonatal sepsis varies between 1 and 8.1 per 1000 live births, although it is lower in developed countries. In our country, the incidence of late-onset sepsis has been reported as 6.4-14.1% and mortality as 0-75%. The incidence of sepsis is 3-10 times higher in preterm babies than in term babies. Disturbances in the establishment of normal intestinal microbiota and commensal microbes colonizing the digestive tract may increase the risk of sepsis through disruption of the mucosal barrier resulting in translocation of luminal contents. Although the correlation of disruptions in the intestinal microbiota with LOS is known, more microbiota-based studies are needed for early intervention to prevent LOS in high-risk infants.

The infant's gut microbiota is a highly dynamic community that is gradually and continuously shaped in the first days of life. Colonization of the infant microbiome begins at birth, when infants can acquire many different types of bacteria from the environment, from their mothers' vagina, skin, and intestines. The immature gut response and changes in the gut microbiota or abnormal colonization pattern in preterm infants predispose the intestines of newborns to inflammation and a range of pro-inflammatory and counter-inflammatory cytokine responses. Microbial translocation or increased permeability to microbial components can then initiate systemic inflammatory response syndrome (SIRS), LOS, NEC, and multisystem organ failure. Native gut microbes are an important source of maturation signals to the infant's developing immune system. Promoting the development of a healthy microbiota in preterm infants is important in preventing NEC and LOS , but the key question is whether natural colonization and succession of microbiota is possible in these infants.

Probiotics are defined as live microorganisms that benefit the host and are often administered enterally to colonize the gastrointestinal tract. Preterm infants are at risk for alterations in the normal protective microbiome due to increased rates of cesarean delivery, exposure to antibiotics, exposure to hospital-acquired pathogens, lack of skin contact with maternal flora, as well as conditions that preclude exposure to breast milk. Modifications of the neonatal microbiome can have long-term effects on health that can last into adulthood. Probiotics are used for various purposes, including preventing NEC and LOS in newborns and infants, reducing the risk of infectious and atopic diseases and treatment duration.

Multiple systematic reviews, meta-analyses, and network meta-analyses examining the results of randomized controlled trials involving more than 10,000 preterm infants have shown significant reductions in NEC and death with probiotic supplementation. When the literature is examined, there are many studies examining prophylactic probiotic supplementation. However, these studies were conducted by giving probiotics directly to babies. Although routine prophylactic probiotic supplementation in preterm infants is controversial, the safety of probiotic supplements is an important issue that should be emphasized. Although there are studies reporting neonatal lactobacillus sepsis,caution is recommended before using probiotics for prophylaxis in immunocompromised patients such as preterms.

Although there are many studies and meta-analyses on the use of probiotics in preterm infants, the purity and numbers of live organisms in the products used, reports of probiotic sepsis and contaminated probiotic products, and the lack of evidence regarding the optimal probiotic strain and dose as well as the methodological differences in these studies. and deficiencies have generated controversy and caused many neonatologists to avoid routine probiotic administration. In many countries, probiotic products are introduced to the market by bypassing the rigor of a drug's approval process in terms of safety, effectiveness, and manufacturing standards and are generally available for use in the dietary supplements category. As a result, currently available probiotics have not undergone drug approval steps and cannot be marketed to treat or prevent diseases in preterm infants, including NEC and LOS. If a probiotic is to be marketed as a drug for the treatment of a disease or disorder, it must meet more stringent requirements, including evidence of safety, efficacy, and approval as a drug for its intended use through clinical trials. The 2010 Clinical Report of the American Academy of Pediatrics, written by the Committee on Nutrition, states that there is insufficient data to recommend probiotics in very low birth weight infants, and because not all probiotics have been studied, not all of them can be generally recommended. The European Committee on Pediatric Gastroenterology, Hepatology and Nutrition recommends caution in administering potentially infectious agents to VLBW babies due to their immunological immaturity, but also states that there is insufficient data to conclude that probiotic administration to preterm newborns is safe. Safety concerns regarding direct administration of probiotics to preterm infants and evidence showing that probiotics given to preterm infants reduce NEC and mortality, support a normal microbiome. has increased interest in alternative methods for safe stimulation. Since it is known that maternal flora and breast milk bacteria are naturally transmitted to fetuses and newborns, an alternative probiotic exposure method that does not directly apply to preterm babies and therefore eliminates the risk of transmission of possible contaminants is the administration of probiotics to mothers of preterm babies.Consumption of breast milk contributes greatly to the colonization of newborn babies (Evidence level: 1 +, Recommendation level: A). Studies have shown that there are more than 200 bacterial species in breast milk, with Lactobacillus and Bifidobacteria predominating, in addition to Staphylococcus , Streptococcus , and Corynebacteria. There is evidence that the neonatal gut microbiome reflects the bacteria found in breast milk and maternal feces. According to the entero-mammary pathway theory, bacteria settle in the breast milk ducts from the mother's gastrointestinal tract through active transport from the blood. Dendritic cells in the maternal intestinal lumen are thought to capture bacteria and transport them to the breast via the blood with the help of mononuclear cells.

Since the human gut has evolved to carry a microbiota, it uses this microbiota to guide developmental cues and various functions. Therefore, shaping the microbiota through breast milk may affect lifelong health. The reduced incidence of NEC and LOS in breast-fed preterm infants is thought to be strictly related to changes in the microbiome. Deoxygenation of the infant gut over time is critical for the acquisition of difficult anaerobes (Bifidobacteria, Bacteroides, Clostridia) that are essential for the healthy function of the microbiome. It has been hypothesized that facultative anaerobes may contribute to deoxygenation, but these organisms are also dangerous to the host. However, how many facultative anaerobes are in the infant intestine, how long they colonize, and how they attach to the infant intestine are clearly regulated by the components of breast milk. Therefore, it seems more reasonable to observe the results by giving probiotics to mothers. The exact mode of action of probiotics is likely strain dependent and difficult to assess due to the overall complexity of the microbiota and interaction with the immune system. In vitro and in vivo studies have shown that Lactobacillus and Bifidobacterium protect the intestinal tract by reducing intestinal permeability and improving intestinal epithelial resistance. exerts direct effects on epithelial barrier function. In our study, mothers in the intervention group will be given 80 ml probiotic product support containing the Actiregularis (5×106 CFU\mL) (lactobacillus bulgaricus, streptococcus thermophilus, lactococcus lactis and bifidobacterium lactis) strain. Although there are a limited number of studies conducted abroad on this subject, as far as we know, our project has a unique value as it is the first project in which stool microbiota results were evaluated in preterm babies by giving probiotics to mothers both in our country and abroad. It carries.

Indirect hyperbilirubinemia in preterm infants is a common phenomenon caused by high bilirubin production due to limited conjugation. Delay in starting enteral feeding in preterm babies, etc. These conditions limit intestinal flow and bacterial colonization, leading to increased enterohepatic circulation of bilirubin. It has been shown that feeding preterm babies supplemented with probiotics regulates gastrointestinal motility and reduces enterohepatic circulation.There are studies showing that the effect of probiotics on the course of hyperbilirubinemia is effective in shortening the duration of phototherapy Another unique value of our project is that probiotic support will be given to mothers and the duration of phototherapy in babies will be evaluated.

Extrauterine growth restriction at discharge is common in preterm infants and is associated with slower growth rates during hospitalization, associated with significant calorie and protein deficiencies and preterm complications.Therefore, optimizing nutrition for preterm infants is among the priority goals. Another effect of probiotic supplementation to preterm babies is a significant decrease in the time to reach full enteral feeding. Other benefits include increased weight gain and reduced time to regain birth weight, shorter hospital stay and fewer episodes of food intolerance, reduced time to transition from orogastric to breastfeeding, and increased postprandial mesenteric flow. In this project, other parameters to be evaluated include the probiotic given to mothers, the baby's weight gain, length of hospital stay, and time to transition to oral feeding.

Breast milk and breastfeeding training will be given by the researcher who has received breast milk and breastfeeding consultancy training in order to ensure that mothers give only breast milk for 20 days, which is one of the criteria for achieving the outcome goals of this project. The fact that breastfeeding consultancy will be provided within the scope of the project is another unique value of the project in terms of protecting and improving mother-child health due to regional characteristics (the province with the highest fertility and child population).

As a result, with this project, the incidence of NEC and LOS in preterm babies due to the use of probiotics added to maternal nutrition, as well as weight gain in babies, duration of phototherapy, time to transition to oral nutrition and hospitalization times will be evaluated. In many studies, probiotics were given to babies and the results were examined. However, the adverse relationship between the safety concerns mentioned above and the current benefits of probiotics leads to the search for a safer route of administration for preterm babies. Although there are a limited number of studies on this subject, the unique value of our project is that probiotic support will be provided to mothers of preterm babies.

Research Hypotheses There is a difference in the incidence of NEC between the intervention and control groups.

There is a difference in the incidence of LOS between the intervention and control groups.

There is a difference between the intervention and control groups in terms of the duration of phototherapy.

There is a difference between the intervention and control groups in terms of time to transition to oral feeding.

There is a difference between the intervention and control groups in terms of growth (weight and head circumference) indicators of babies.

There is a difference in length of hospital stay between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Mothers;

* Being 18 years or older
* Having the ability to read, write and understand Turkish,
* Having a singleton pregnancy,
* Birth time is between 28-32 weeks of gestation,
* Not being a smoker
* Being able to breastfeed your baby at least 8-10 times a day
* The mother does not have any diagnosed digestive system disease (ulcerative colitis, Crohn's disease, etc.) (This information will be obtained from the mother's file)
* Volunteering to participate in the research

Inclusion Criteria for Babies:

• The baby's gestational age is between 28-32 weeks (including the 28th and 32nd weeks)

Exclusion Criteria:

Exclusion Criteria for Mothers from the Study;

* The mother has problems with expressing milk or breast problems,
* The mother has a chronic disease (pre-existing clinical conditions such as diabetes, hypertension, hypothyroidism, autoimmune diseases, asthma, allergy, kidney or liver diseases, viral, bacterial or protozoan infection, anemia (hemoglobin, Hb<0 g/L), etc.). to be
* The mother is using another probiotic product
* The mother does not use the recommended probiotic appropriately and at the appropriate time.
* Giving breast milk to the baby less than 8 times for 2 consecutive days,
* The sampled mother is also included in other clinical studies.

Exclusion Criteria for Babies from the Study;

* The baby uses formula other than breast milk for more than 24 hours
* The baby has a health problem that prevents breastfeeding
* Presence of genetic and metabolic disease in the baby,
* Congenital anomaly in the baby,
* Presence of neurological, gastrointestinal or major cardiac anomalies and/or hypoxic brain damage.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Necrotizan Enterocolit (NEC) | 4 months
  Preterm baby diagnosed with NEC(Whether or not NEC was diagnosed as stage 2 or higher according to Bell staging)
Late Onset Sepsis(LOS) | 4 months
  Preterm baby diagnosed with LOS(whether they have been diagnosed with sepsis confirmed by a positive blood culture
head circumference measurement | 4 months
  head circumference measurement of preterm baby(Change in head circumference to be measured weekly (in centimeters))
weight measurement of preterm baby | 4 months
  Weight measurement of the premature baby (weight measurement will be measured weekly (in grams))
Hyperbilirubinemia | 4 months
  measuring total bilirubin level on the 1st and 5th day of birth
Phototherapy | 4 months
  How many hours of phototherapy the baby received during hospitalization
Full oral Feeding | 4 months
  Time for the preterm baby to transition to full oral feeding
Hospitalization Day | 4 months
  Hospitalization period (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Alev Esercan, Study Chair — https://sanliurfaeah.saglik.gov.tr/

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to be shared when the study is completed and published.